CLINICAL TRIAL: NCT07371260
Title: Effects of Virtual Reality With Multisensory Stimulation on Emotional and Behavioral Disorders in Individuals With Acquired Brain Injury and Disability Requiring Institutional Care: a Single Case Experimental Design (SCED) Study.
Acronym: Rév In MAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Musse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A02119-40
Record Dates: First submitted 2026-01-09; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Brain Injury; Virtual Reality; Behavior; Emotion; Well-being
Keywords: Acquired Brain Injury; Behavior; Emotion; Well-being; Virtual Reality; Multisensory; Specialized Care Home
MeSH Terms: conditions — Brain Injuries; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): VR
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — The intervention will consist of 8 weeks with two weekly virtual relaxation sessions using the VirtySens® multisensory device, lasting 15 to 20 minutes.

SUMMARY:
Acquired brain injuries (ABIs) frequently cause emotional and behavioral disorders that impair independence and quality of life, particularly in institutions. Virtual reality (VR), already used in various mental and neurological disorders, offers therapeutic potential that remains largely unexplored in this context.

Multisensory devices offer enhanced immersion that can potentially increase the relaxation and calming effect. Their use in specialized care home (SCH) could provide additional support for care.

The main objective of the study is to measure the effect of an 8-week multisensory VR relaxation program on the most significant emotional and behavioral disorders in adults with acquired brain injury living in SCH. The SCED method with multiple baselines across subjects (ABA) is used with three adult residents with ABCI and behavioral disorders living in SCH. The study consists of three phases (baseline, intervention, follow-up), during which the three main emotional and behavioral disorders of each resident are assessed weekly based on observations made throughout the week. Additional measures include the assessment of the socio-emotional profile by the care team (ECCSEG) and the emotional distress experienced by residents (QOLIBRI), collected twice per phase. The intervention consists of eight weeks of VR relaxation (VirtySens®), with two 15-minute sessions per week.

All measurements taken during the experiment will be anonymized and used only by the investigators, who are fully aware of the European GDPR (General Data Protection Regulation) concerning the protection of personal data.

ELIGIBILITY:
Inclusion Criteria:

* Resident aged over 18
* Diagnosis of stroke, traumatic brain injury, tumor, or cerebral anoxia for more than 3 years.
* Living in a nursing home for at least 6 months
* Presence of one or more emotional and behavioral disorders during initial assessments (NPI-ES) for at least 3 months.
* Sufficient cognitive abilities to understand instructions and answer questions using a Likert scale.
* Normal or corrected visual acuity
* Resident affiliated with the social security system

Exclusion Criteria:

* Motor or sensory disorders incompatible with the use of VR
* Unstabilized photosensitive epilepsy or presence of a seizure in the past year
* Change in the prescription of neuroleptic treatments, antidepressants, benzodiazepines, sedatives, anxiolytics, mood stabilizers, antiepileptics, or betablockers within the last 3 months.
* Unstabilized major psychiatric disorders.
* Craniectomy
* Limited range of cervical movement due to orthopedic disorders
* Moderate or severe hearing loss not compensated by a hearing aid
* Anosmia
* Asthma
* Pregnant women or women suspected of being pregnant
* Breastfeeding women
* Neurocognitive disorders preventing understanding of instructions during assessments
* The resident is included in another research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
NPI-ES | Twice a week, for 21 weeks
  The primary outcome measure is the weekly NPI-ES score, calculated for the three most prominent emotional and behavioral disturbances in each participant.
  This score is calculated from systematic observations made daily over five consecutive days, during two standardized periods of the day: (1) lunch and (2) a group activity in the afternoon.

SECONDARY OUTCOMES:
ECCSEG : The Geneva Scale of Socio-Emotional Behavior Changes | in the middle and at the end of each phase of the SCED (baseline, intervention, follow-up). 6 evaluations
  The Geneva Socio-Emotional Behavior Change Scale (ECCSEG) was developed by Beni et al. (2017) to assess socio-emotional disorders frequently encountered after a TBI, although it can also be used in other etiological contexts. The ECCSEG questionnaire is completed by the neuropsychologist together with the care team, which includes at least one registered nurse, one nursing assistant or medical-psychological assistant, one special education teacher, and one psychomotor therapist during weekly team meetings. The team agrees to evaluate the 22 items on each participant's questionnaire. A total score is then calculated by adding up all the scores per item. The ECCSEG questionnaire is completed twice per phase: midway through and at the end of the phase.
The QOLIBRI Emotion Questionnaire | Twice at baseline, twice during the intervention, and twice during follow-up (6 evaluations).
  The QOLIBRI Emotion Questionnaire is a tool specifically designed for people with brain injuries, which aims to gather subjective perceptions of patients' quality of life.
Sensory capsule satisfaction survey | Twice during the intervention
  Each resident is asked:
  "Are you satisfied with using the sensory capsule? On a scale of 1 to 5 (Likert). 1 = Not at all; 2 = A little; 3 = Moderately; 4 = Quite a lot; 5 = Very much." Why? Residents will answer this question twice during the intervention.
The Simulator Sickness Questionnaire (SSQ) | Twice during the intervention
  The Simulator Sickness Questionnaire (SSQ) is currently the gold standard test for objectively measuring cybersickness.
The RV Presence Questionnaire | Twice during the intervention
  The Presence Questionnaire (74): consisting of 19 items on a 7-point scale, it measures the feeling of presence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: No